CLINICAL TRIAL: NCT07329322
Title: A Randomized, Open-label, Multicenter, Phase II Clinical Study to Evaluate the Safety and Efficacy of Sacituzumab Tirumotecan in Combination With Osimertinib or as Monotherapy for Neoadjuvant Treatment in Patients With Resectable Epidermal Growth Factor Receptor (EGFR)-Mutated Non-Small Cell Lung Cancer
Brief Title: Phase II Study of Sacituzumab Tirumotecan in Combination With Osimertinib or Sacituzumab Tirumotecan for Neoadjuvant Treatment in Patients With Resectable Epidermal Growth Factor Receptor (EGFR)-Mutated Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-II-18
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Tirumotecan+Osimertinib (Experimental): Participants will receive Sacituzumab Tirumotecan for each 2-week cycle, Osimertinib once-daily for each 2-week cycle.
  Interventions: Drug: Sacituzumab Tirumotecan; Drug: Osimertinib
- Sacituzumab Tirumotecan (Experimental): Participants will receive Sacituzumab Tirumotecan for each 2-week cycle
  Interventions: Drug: Sacituzumab Tirumotecan

INTERVENTIONS:
Drug: Sacituzumab Tirumotecan — Sacituzumab Tirumotecan: 4mg/kg, intravenous (IV) infusion
Drug: Osimertinib — 80mg, QD
  Arms: Sacituzumab Tirumotecan+Osimertinib

SUMMARY:
The aim of the study to evaluate the safety and efficacy of Sacituzumab Tirumotecan in combination with osimertinib or as monotherapy for neoadjuvant treatment in patients with resectable Epidermal Growth Factor Receptor (EGFR)-Mutated Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, Phase 2 study to evaluate the safety and efficacy of Sacituzumab Tirumotecan in combination with osimertinib or as monotherapy for neoadjuvant treatment in patients with resectable Epidermal Growth Factor Receptor (EGFR)-Mutated Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 18 and ≤ 75 years at the time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed NSCLC.
3. No prior systemic anti-tumor therapy.
4. No prior local therapy for NSCLC.
5. Confirmed by tumor histology, or cytology to have EGFR sensitizing mutations.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before randomization.
7. At least one target lesion as assessed by the investigator according to RECIST v1.1.
8. Life expectancy ≥ 24 weeks.
9. Adequate organ and bone marrow function.
10. For female participants of childbearing potential and male participants with partners of childbearing potential, they must agree to use effective medical contraception from the start of signing the ICF until 6 months after the last dose.
11. Participants must voluntarily join this study, sign the ICF, and be able to comply with the protocol-specified visits and related procedures.

Exclusion Criteria:

1. Tumor histology or cytology confirming combined small cell lung cancer, neuroendocrine carcinoma, or carcinosarcoma or squamous cell carcinoma components of more than 10%.
2. Participants with other malignant tumors within 3 years prior to randomization.
3. Resting electrocardiogram (ECG) showing clinically significant abnormal results.
4. Presence of any of the following cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors.
5. Uncontrolled systemic diseases in the investigator's judgment.
6. History of interstitial lung disease (ILD), drug-induced ILD, or non-infectious pneumonitis, have current ILD or non-infectious pneumonitis.
7. Clinically severe lung damage due to complications of lung disorder.
8. Participants who have received systemic corticosteroids therapy with > 10 mg/day of prednisone or other immunosuppressive drugs within 2 weeks before randomization.
9. Known active pulmonary tuberculosis.
10. Known history of allogeneic organ transplant and allogeneic hematopoietic stem cell transplant.
11. Active hepatitis B.
12. Positive for human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
13. Known hypersensitivity to osimertinib, sacituzumab tirumotecan, or any of their components (including but not limited to polysorbate-20); known history of severe hypersensitivity to other biologics.
14. Have received a live vaccine within 30 days prior to randomization, or plan to receive a live vaccine during the study.
15. Pregnant or lactating women.
16. Any condition that, in the investigator's opinion, would interfere with the evaluation of the study drug, participant safety, or interpretation of study results, or any other condition that the investigator considers unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) rate | up to 60 months
  MPR rate is defined as the proportion of participants achieving ≤ 10% residual viable tumor cells in the postoperative surgical specimen.

SECONDARY OUTCOMES:
pathological Complete Response (pCR) rate | up to 60 months
  pCR rate is defined as the proportion of participants achieving absence of any residual viable tumor cells in the postoperative surgical specimen.
Residual viable tumor percentage (RVT%) | up to 60 months
  RVT% is defined as the proportion of residual viable tumor cells in the postoperative surgical specimen.
R0 resection rate | up to 60 months
  Proportion of participants achieving R0 resection
Pathological lymph node downstaging rate | up to 60 months
  Pathological lymph node downstaging rate is defined as the proportion of participants achieving pathological lymph node downstaging
Pathological primary tumor downstaging rate | up to 60 months
  Pathological primary tumor downstaging rate is defined as the proportion of participants achieving pathological primary tumor downstaging
ORR | up to 60 months
  ORR is defined as a partial or complete response according to RECIST, version 1.1.
EFS | up to 60 months
  EFS is defined as the time from randomization to progression of disease, recurrence of disease, or death from any cause.
DFS | up to 60 months
  DFS is defined as the time from surgery to disease progression (recurrence or metastasis) or death due to any cause.
OS | up to 60 moths
  OS is defined as the time from randomization to death from any cause.
Incidence of Adverse events (AEs) and serious adverse events (SAEs) as assessed by NCI CTCAE v5.0 | up to 60 months
  Incidence (based on NCI CTCAE v5.0) of adverse events (AEs) and serious adverse events (SAEs).
Severity of Adverse events (AEs) and serious adverse events (SAEs) as assessed by NCI CTCAE v5.0 | up to 60 months
  Severity (based on NCI CTCAE v5.0) of adverse events (AEs) and serious adverse events (SAEs).
Maximum observed plasma concentration (Cmax) of Sacituzumab Tirumotecan-ADC, Sacituzumab Tirumotecan-TAB, and free KL610023 | up to 60 months
  To assess the pharmacokinetic (PK) profile of Sacituzumab Tirumotecan.
Anti-drug Antibodies (ADA) of Sacituzumab Tirumotecan | up to 60 months
  Immunogenicity test results of Sacituzumab Tirumotecan.